CLINICAL TRIAL: NCT04875715
Title: Prospective Evaluation of Topical Almond Oil vs Hydroquinone on the Appearance of Facial Pigmentation and the Stability of the Microbiome
Brief Title: Prospective Evaluation of Topical Almond Oil vs Hydroquinone
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 1666478
Record Dates: First submitted 2021-03-05; First posted 2021-05-06 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Skin Pigmentation
MeSH Terms: conditions — Pigmentation Disorders | interventions — almond oil; hydroquinone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Almond oil (Experimental): Almond Oil Pressed Cold
  Interventions: Other: Almond Oil
- Hydroquinone (Active Comparator): Hydroquinone 2% cream
  Interventions: Drug: Hydroquinone Topical

INTERVENTIONS:
Other: Almond Oil — Almond oil
  Arms: Almond oil
Drug: Hydroquinone Topical — Hydroquinone 2% cream
  Other Names: Hydroquinone
  Arms: Hydroquinone

SUMMARY:
The purpose of this study is to analyze facial pigmentation and skin microbiome changes after topical almond oil application, compared to the use of topical hydroquinone.

DETAILED DESCRIPTION:
The purpose of this experiment is to analyze facial pigmentation and skin microbiome changes after topical almond oil application, compared to the use of topical hydroquinone.

There will be a total of 50 subjects:

* 25 randomized to receive almond oil nightly
* 25 randomized to receive 2% hydroquinone nightly

Study Timelines:

* The duration of an individual subject's participation will last from the day of the consent/screening (visit 1) until visit 5 where they will have images taken and measurements collected to assess skin pigment, skin hydration, sebum excretion rate.
* The duration of participation is 4 months.
* The estimated time for the investigators to complete primary analysis is 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal women of Fitzpatrick skin types 3 to 6

Exclusion Criteria:

* Those with a nut allergy
* Smoking is an independent risk factor and serves as a confounder for the development of facial aging [18]. Therefore current smokers, those that have smoked within the past year, and former smokers with greater than a 20 pack year history of smoking will be excluded.
* Those with an autoimmune photosensitive condition or a known genetic condition with a deficiency in collagen production (such as Ehlers-Danlos syndrome) will be excluded as this can be a confounder for facial photoaging.
* Hormonal medications or therapies will not be allowed unless they have been stable on their medications for at least 2 months. Examples include oral contraceptives, progesterone-based injections, and estrogen based hormonal replacement therapy.
* Those who have undergone any cosmetic procedures to the face in the 4 months prior to enrollment in the opinion of the investigator. People that have undergone deeper chemical peels (TCA based peels) within 1 year prior to enrollment will also not be eligible.
* Individuals who are unwilling to discontinue vitamin E containing supplements and food sources during the washout and intervention.
* Individual who are unwilling to discontinue topical cosmetic products during the duration of the study.
* Individuals who are not willing to engage in a two-week washout on topical treatments known to affect facial pigmentation and these agents will be restricted during the study period as well. These include topicals that contain:

  * Retinoids such as tretinoin, adapalene, retinol.
  * Antioxidant ingredients such as vitamin C or vitamin E.
  * Pigment-reducing agents such as hydroquinone, azelaic acid, kojic acid per the discretion of the investigator except for the hydroquinone that is provided in this study.
  * Topicals that contain a nut oil or nut extract as part of their ingredient list.
* Furthermore, subjects will be asked to refrain from use of any other topical products for one week prior to each visit apart from the study agents supplied from this study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Premenopausal women
Enrollment: 50 (Estimated)
Dates: Start 2021-07-01 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Intensity of facial pigment | 16 weeks
  Facial images will be obtained and analyzed with the BTBP image analysis system

SECONDARY OUTCOMES:
Shifts in the microbiome diversity (Shannon index as an example) | 16 weeks
  The skin microbiome will be analyzed to assess any changes after topical almond oil application, compared to the use of topical hydroquinone.
Quantification for the presence of species within the genus Cutibacteria, Staphyloccoccus, and Ralstonia | 16 weeks
  The skin microbiome will be analyzed to assess the presence of species within the genus Cutibacteria, Staphyloccoccus, and Ralstonia
Appearance of facial redness | 16 weeks
  The research team will quantify the presence of facial redness with a SkinColorCatch from Delfin Technologies. This will measure the RGB colors and average them from each participant for each of the visits.
  Skin pigment, including the presence of redness, will be measured using a SkinColorCatch from Delfin Technologies. This device shows the RGB Colors, CIE L*a*b* and L*c*h* color space coordinates when the device is applied to the skin.Included is the link to the device (http://www.truesystem.co.kr/product/pdf/SkinColorCatch%20Brochure%202016.pdf).
Subjective tolerability assessment | 16 weeks
  A questionnaire that assesses for stinging, itching, and burning will be utilized.
Intensity of facial pigment | 8 weeks
  Facial images will be obtained and analyzed with the BTBP image analysis system

CONTACTS AND LOCATIONS:
Overall Officials: Raja Sivamani, MD MS AP, Principal Investigator — UC Davis Dermatology
Locations (1):
- UC Davis Department of Dermatology, Clinical Trials Unit, Sacramento, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Learn more or sign up for the study here! — https://studypages.com/s/prospective-evaluation-of-topical-almond-oil-vs-hydroquinone-336267/